CLINICAL TRIAL: NCT02082782
Title: Colorectal Metastatic Liver Disease: Efficacy of Irreversible Electroporation (IRE) - a Phase II Clinical Trial (COLDFIRE-2 Study)
Brief Title: Efficacy of Irreversible Electroporation (IRE) for Central Colorectal Liver Metastases
Acronym: COLDFIRE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. M.R. Meijerink, Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLDFIRE-2 study
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal liver metastases (CRLM); Tumor ablation; Irreversible electroporation (IRE); Interventional oncology; NanoKnife; Colorectal liver metastasis, unresectable and not-thermally ablative due to location near vulnerable structures like vessels or bile ducts
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: Single arm prospective trial with predefined endpoint: accept indication if at least 50% of patients are alive without local tumor progression at 12 months following irreversible electroporation (IRE) treatment for centrally located colorectal cancer liver metastases (CRLM)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irreversible electroporation (IRE) (Experimental): Single arm study: percutaneous or open irreversible electropration of CRLM
  Interventions: Procedure: Irreversible electroporation (IRE)

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE) — Percutaneous (CT-guided) or open (US-guided) irreversible electroporation of central colorectal liver metastasis.
  Other Names: NanoKnife

SUMMARY:
Irreversible electroporation (IRE) is a new, minimal-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels and bile ducts. With IRE, multiple electrical pulses are applied to tumorous tissue. These pulses alter the existing transmembrane potential of the cell membranes, and create 'nanopores', after which the cell dies through loss of homeastasis.

The purpose of this study is to investigate the efficacy of percutaneous and open IRE in the treatment of patients with colorectal liver metastases (CRLM) that are unsuitable for resection or thermal ablation due to vicinity to vulnerable structures such as vessels and bile ducts. Other objectives are safety, feasibility (technical success) and imaging characteristics on follow-up (PET-)CT and PET-MRI and the value of these imaging modalities in dianosing local site recurrence (LSR) or residual disease (RD).

29 patients with histologically confirmed colorectal carcinoma who present with unresectable and not thermally ablative CRLM< 3.5cm suitable for IRE will undergo percutaneous or open irreversible electroporation of the tumor using CT and ultrasound guidance. All (serious) adverse events are registered. One day post-IRE MRI is performed to assess technical success. Follow-up will consist of frequent (PET-)CT and (PET-)MRI scanning to localize residual or recurrent disease. Overall technique effectiveness is determined 1 year after treatment.

The investigators hypothesize that IRE for central CRLM will lead to good tumor control without causing severe complications.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of primary colorectal tumor;
* Previous induction chemotherapy due to unresectability; no intra- or extrahepatic disease progression under induction chemotherapy; OR
* Previous chemotherapy for other CRLM, now presenting with renewed CRLM unsuitable for resection or thermal ablation;
* Liver metastases F-18-FDG PET avid and visible on ceCT, size ≤ 3,5 cm and not eligible for resection or thermal ablation due to location close to a vessel or bile duct;
* Age more than 18 years;
* ASA classification 0 - 3;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to definite inclusion:

  * Hemoglobin ≥ 5.6 mmol/L;
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3;
  * Platelet count ≥ 100*109/l;
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * ALT and AST ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance > 50 ml/min;
  * Prothrombin time or INR < 1.5 x ULN;
  * Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed if this treatment can be interrupted as judged by the treating physician)
* Written informed consent

Exclusion Criteria:

* Lesion > 3,5 cm size;
* History of epilepsy;
* Extrahepatic metastases rendering local therapy unfeasible;
* History of cardiac disease:

  * Congestive heart failure >NYHA class 2;
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening);
  * Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers are permitted);
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Pregnant or breast-feeding subjects;
* Immunotherapy ≤ 6 weeks prior to the procedure;
* Chemotherapy ≤ 6 weeks prior to the procedure;
* Concomitant use of anti-convulsives and anti-arrhythmic drugs other than beta blockers for antiepileptic or antiarrhythmic purpose;
* Allergy to contrast media;
* Any implanted stimulation device;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 months
  The primary objective of this project is to evaluate the efficacy (percentage of lesions that show no sign of recurrence 12 months after the initail IRE procedure) of IRE for CRLM on cross-sectional imaging performed after respectively 6 weeks, and after 3, 6, 9 and 12 months. Research has shown that 95% of all recurrences after RFA of CRLM are diagnosed within one year after treatment. Therefore, one year follow-up will allow for accurate calculation of efficacy. Exact secondary efficacy rate may require follow-up longer than 12 months since this includes lesions that have been re-treated due to local site recurrence/local tumor residue (which will be individualized for each patient after re-treatment of LSR/LTR).

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R Meijerink, MD, PhD, Principal Investigator — VU University Medical Center (VUmc); Krijn P van Lienden, MD, PhD, Principal Investigator — Academic Medical Center Amsterdam (AMC); Arian R van Erkel, MD, PhD, Principal Investigator — Leiden University Medical Center (LUMC)
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland

REFERENCES:
- [Derived] Meijerink MR, Ruarus AH, Vroomen LGPH, Puijk RS, Geboers B, Nieuwenhuizen S, van den Bemd BAT, Nielsen K, de Vries JJJ, van Lienden KP, Lissenberg-Witte BI, van den Tol MP, Scheffer HJ. Irreversible Electroporation to Treat Unresectable Colorectal Liver Metastases (COLDFIRE-2): A Phase II, Two-Center, Single-Arm Clinical Trial. Radiology. 2021 May;299(2):470-480. doi: 10.1148/radiol.2021203089. Epub 2021 Mar 16. PMID 33724066
- [Derived] Scheffer HJ, Vroomen LG, Nielsen K, van Tilborg AA, Comans EF, van Kuijk C, van der Meijs BB, van den Bergh J, van den Tol PM, Meijerink MR. Colorectal liver metastatic disease: efficacy of irreversible electroporation--a single-arm phase II clinical trial (COLDFIRE-2 trial). BMC Cancer. 2015 Oct 24;15:772. doi: 10.1186/s12885-015-1736-5. PMID 26497813